CLINICAL TRIAL: NCT03171987
Title: The Safety and Efficacy of 5% Lidocaine Patch and Flurbiprofen Patch for Relieving Acute Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Principal Investigator, Meng-Huang Wu, Orthopedic specialist, Taipei Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N201702048
Record Dates: First submitted 2017-05-24; First posted 2017-05-31 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2021-03

CONDITIONS: Acute Back Pain
Keywords: lidocaine patch; flurbiprofen patch; acute back pain

STUDY DESIGN:
Intervention Model Description: 1. Lidocaine patch group: 1 piece lidocaine patch per day at back pain area. The treatment lasts for 28 days.
  2. Flurbiprofen patch group: 1 piece flurbiprofen patch per day at back pain area. The treatment lasts for 28 days.
Who Masked: Care Provider, Investigator
Masking Description: The investigator and care provider will be blind to group. Participant will know their treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine patch (Experimental): Lidocaine patch local application 1 piece per day for 28 days at back pain area.
  Interventions: Drug: Lidocaine patch local application
- Flurbiprofen patch (Active Comparator): Flurbiprofen patch local application 1 piece per day for 28 days at back pain area.
  Interventions: Drug: Flurbiprofen patch local application

INTERVENTIONS:
Drug: Lidocaine patch local application — Attach the patch to back pain area 1 piece per day with no more than 6 hours.
  Other Names: Lidopat patch
  Arms: Lidocaine patch
Drug: Flurbiprofen patch local application — Attach the patch to back pain area 1 piece per day with no more than 6 hours.
  Arms: Flurbiprofen patch

SUMMARY:
This is a prospective, randomized, single blinded, two-arm, head to head study.

The purpose of this study is:

* To evaluate and compare the efficacy of 5% lidocaine patch and flurbiprofen patch for treatment of acute low back pain.

Determining the effect of the 5% lidocaine patch and flurbiprofen patch for improving functional disabilities and in reducing pain resulting from acute low back pain. Efficacy will be determined by the level of pain relief (as measured by the Numerical Rating Scale, NRS), decrease in analgesics, improved quality of life (as measured by the Oswestry Disability Questionnaire, ODQ, and core outcome measures index questionnaire, COMI), pain interference with function (as measured by the Brief Pain Inventory-Interference scale, BPI-QoL), Short-Form McGill Pain Questionnaire-2(SF-MPQ-2), general health status (as measured by the EQ5D), Overall treatment effect (OTE), physical exam from baseline up to 1-Months.

ELIGIBILITY:
Inclusion Criteria:

* All subjects underwent a detailed history and systemic physical examination including neurologic and musculoskeletal evaluations. To rule out any confounding etiologies, basic diagnostic laboratory tests including complete blood count and acute phase reactants (erythrocyte sedimentation rate and C-reactive protein) were performed. The patients diagnosed as having acute non-specific low back pain according to history and physical examinations were invited to participate and will be informed about the purpose and course of the study.

Main inclusion criteria

* A primary complaint of pain in the area between the 12th rib and buttock crease without leg pain
* Female or male, 20 - 80 years of age
* Low back pain of less than six weeks' duration; and at least moderate pain intensity (NRS≧4)

Exclusion Criteria:

Main exclusion criteria:

* Known or suspected serious spinal pathology and spinal implants
* Lumbar spinal surgery within the preceding six months
* Serious comorbidities preventing prescription of paracetamol
* Alternative treatment for low back pain in previous two weeks
* Chronic neurological lesion
* Chronic musculoskeletal lesion
* Active cancer
* Pregnancy
* Use of pain medication (except paracetamol) within 3 days
* Treatment site has active skin lesion or inflammation
* Known allergy to skin patch

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) | 28 day
  Back pain relief effectiveness

SECONDARY OUTCOMES:
Numeric rating scale (NRS) | 0, 1, 3, 7, 14, 21 day
  Back pain relief effectiveness
Brief Pain Inventory-Quality of Life (BPI-QoL) | 0, 7, 14, 21, 28 day
  Back pain relief effectiveness
Oswestry Disability Questionnaire (ODQ) | 0, 7, 14, 21, 28 day
  Back pain relief effectiveness
Core Outcome Measurement Index (COMI) | 0, 7, 14, 21, 28 day
  Back pain relief effectiveness
EQ5D Quality of Life questionnaires Efficacy | 0, 7, 14, 21, 28 day
  Back pain relief effectiveness
Short form-Mcgill Pain Questionnaire (SF-MPQ-2) | 0, 7, 14, 21, 28 day
  Back pain relief effectiveness
Overall Treatment Effect Scale (OTE) | 7, 14, 21, 28 day
  Back pain relief effectiveness
Analgesic consumption | 7, 14, 21, 28 day
  Back pain relief effectiveness
Skin reaction grade (Assessment of dermal response) | 1, 3, 7, 14, 21, 28 days
  Safety
Common Terminology Criteria for Adverse Events (CTCAE) | 1, 3, 7, 14, 21, 28 days
  Safety

OTHER OUTCOMES:
Physical exams for back range of motion | 0, 7, 14, 21, 28 day
  Back pain relief effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Ray-Jade Chen, MD, Study Chair — Taipei Medical University Hospital
Locations (2):
- Taiwan (2):
  - Postal Hospital, Taipei
  - Taipei Medical University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No
No shore IPD plan.

REFERENCES:
- [Background] Coste J, Lefrancois G, Guillemin F, Pouchot J; French Study Group for Quality of Life in Rheumatology. Prognosis and quality of life in patients with acute low back pain: insights from a comprehensive inception cohort study. Arthritis Rheum. 2004 Apr 15;51(2):168-76. doi: 10.1002/art.20235. PMID 15077256
- [Background] Mick G, Correa-Illanes G. Topical pain management with the 5% lidocaine medicated plaster--a review. Curr Med Res Opin. 2012 Jun;28(6):937-51. doi: 10.1185/03007995.2012.690339. Epub 2012 May 24. PMID 22551228
- [Background] Bolten W. The pharmacokinetics, pharmacodynamics and comparative efficacy of flurbiprofen LAT. Br J Clin Pract. 1994 Jul-Aug;48(4):190-5. PMID 7917798